CLINICAL TRIAL: NCT04567316
Title: A Phase I, Open-label Trial to Investigate Metabolism and Pharmacokinetics of a Single Dose of [14C] BI 1358894 Administered as Oral Solution (Part 1) and Multiple Doses of BI 1358894 Administered as Film-coated Tablets (Part 2) in Healthy Male Volunteers
Brief Title: A Study in Healthy Men to Test How BI 1358894 is Taken up and Handled by the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1402-0015; 2020-002054-25 (EudraCT Number)
Record Dates: First submitted 2020-09-25; First posted 2020-09-28 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — TRPC inhibitor BI 1358894

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- [14C]-radiolabelled BI 1358894 (Experimental): [14C]-radiolabelled BI 1358894 (part 1)
  Interventions: Drug: [14C]-radiolabelled BI 1358894
- BI 1358894 (Experimental): BI 1358894 (part 2)
  Interventions: Drug: BI 1358894

INTERVENTIONS:
Drug: [14C]-radiolabelled BI 1358894 — Part 1
  Arms: [14C]-radiolabelled BI 1358894
Drug: BI 1358894 — Part 2
  Arms: BI 1358894

SUMMARY:
The main objective of this trial is to investigate the basic pharmacokinetics of BI 1358894 and its metabolites, total radioactivity, including mass balance, excretion pathways and metabolism following a single oral dose of [14C] BI 1358894 in Part 1 and to investigate the pharmacokinetics of BI 1358894 and its metabolite(s) following multiple-dose treatment over 21 days with non- radiolabelled compound of BI 1358894 in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 65 years (inclusive)
* BMI of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation
* Male subjects who meet any of the following criteria from screening until 90 days after trial completion:

  * Use of adequate contraception of the female partner, e.g. any of the following methods plus condom: implants, injectables, combined oral or vaginal contraceptives, intrauterine device that started at least two months prior to first study drug administration or barrier method (e.g. diaphragm with spermicide) or,
  * Sexually abstinent or,
  * A vasectomy performed at least 1 year prior to screening (with medical assessment of the surgical success) or,
  * Surgically sterilised female partner (including hysterectomy, bilateral tubal occlusion, or bilateral oophorectomy) or,
  * Postmenopausal female partner, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with levels of follicle-stimulating Hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 40 to 100 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* C-reactive protein (CRP) > upper limit of normal (ULN), liver or kidney parameter above ULN
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* For Part 1 only:

  * Participation in another absorption, distribution, metabolism, and excretion (ADME) pharmacokinetics study with a radiation burden of >0.1 millisievert (mSv) in the period of 1 year prior to screening
  * Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton (excluding spinal column)) in the period of 1 year prior to screening
  * Irregular defecation pattern (less than a mean of one bowel movement every 1 or 2 days)

In addition, the following Severe acute respiratory syndrome coronavirus type 2 (SARS-CoV-2) specific exclusion criterion apply:

* A positive test indicating an ongoing infection with SARS-CoV-2 and clinical symptoms suggestive of the disease
* Further exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-01-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ICON, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a phase I, open-label trial to investigate metabolism and pharmacokinetics of a single dose of [14C] BI 1358894 administered as oral solution (Part1) and multiple doses of BI 1358894 administered as film-coated tablets (Part 2) in healthy male volunteers.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- 100 mg [14C]-Radiolabeled BI 1358894 (Part 1): Single dose (SD) of 100 milligram (mg) of radiolabeled BI 1358894 was administered as oral solution on Day 1. Oral solution contained a mixture of Carbon 14-radiolabelled BI 1358894 ([14C] BI 1358894) corresponding to a radioactive dose of 3.7 megabecquerels (MBq) (100 microcuries (μCi)) in a solution of 10 milliliter (mL) volume (concentration of BI 1358894 10 mg/mL).
- 100 mg BI 1358894 (Part 2): Multiple doses (MD) of 2 non-radiolabeled film-coated tablets of 50 milligram (mg) BI 1358894 were administered orally once daily (QD) from Day 1 to Day 21 with 240 milliliter (mL) of water .
Period: Overall Study
Arm/Group | 100 mg [14C]-Radiolabeled BI 1358894 (Part 1) | 100 mg BI 1358894 (Part 2)
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This subject set included all subjects who entered the study who were documented to have received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 mg [14C]-Radiolabeled BI 1358894 (Part 1) | 100 mg BI 1358894 (Part 2) | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.4 (19.2) | 39.1 (20.0) | 40.3 (18.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Mass Balance and Recoveries of [14C] BI 1358894 Total Radioactivity in Urine and Faeces After Single Oral Dose (Fe0-tz)
Description: Mass balance and recoveries of [14C] BI 1358894 total radioactivity in urine and faeces after single oral dose as percentage of the administered dose over the time interval from 0 to tz, where tz is the latest quantifiable data point across all participants.
  Urine collection intervals were within 2 hours (h) predose, 0-4, 4-8, 8-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216, 216-240, 240-264, 264-288, 288-312, 312-336 h after dosing on Day 1 and to be continued in 24 h intervals, on days 21-22, 28-29, 35-36, 42-43, and 49-50, if necessary.
  Faeces collection intervals were started from approximately -48 h before drug administration and 0-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216, 216-240, 240-264, 264-288, 288-312, 312-336 h after dosing on Day 1 and to be continued in 24 h intervals, on days 21-22, 28-29, 35-36, 42-43, and 49-50, if necessary.
Time Frame: From within 2 hours predose up to 50 days after dosing. For detailed time frames please refer to the intervals given under "measure description" above.
Population: Pharmacokinetic set (PKS) Part 1: This subject set included all subjects in treated set (TS) who provided at least one primary or secondary PK parameter that was not excluded according to description above. Thus, a subject was included in PKS, even if he/she contributed only one pharmacokinetics (PK) parameter value to the statistical assessment. Only subjects with available data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of administered dose
Arm/Group | 100 mg [14C]-Radiolabeled BI 1358894 (Part 1)
Number analyzed (Participants) | 7
Percentage of administered dose | 85.8 (3.42)

2. Secondary Outcome: Part 1: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) were determined for total [14C] BI 1358894 and non-radiolabeled BI 1358894 after single dose administration.
Time Frame: At 2 hours (h) before first drug administration and at 20 minutes (min), 40min, 1h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 36h, 48h, 72h, 96h, 120h, 144h, 192h, 240h, 288h, 336h, 485h, 653h after first drug administration.
Population: Pharmacokinetic set (PKS) Part 1: This subject set included all subjects in the TS who provided at least one primary or secondary PK parameter that was not excluded according to the description above. Thus, a subject was included in the PKS, even if he/she contributed only one PK parameter value to the statistical assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours * nanomol / Liter
Arm/Group | 100 mg [14C]-Radiolabeled BI 1358894 (Part 1)
Number analyzed (Participants) | 8
Hours * nanomol / Liter
  BI 1358894 | 13000 (30.9)
  [14C] BI 1358894-EQ | 73200 (26.8)

3. Secondary Outcome: Part 1: Maximum Measured Concentration of the Analyte in Plasma (Cmax)
Description: Maximum measured concentration of the analyte in plasma (Cmax) determined for total [14C] BI 1358894 and non-radiolabeled BI 1358894 after single dose administration.
Time Frame: as for outcome 2
Population: Pharmacokinetic set (PKS): This subject set included all subjects in the TS who provided at least one primary or secondary PK parameter that was not excluded according to the description above. Thus, a subject was included in the PKS, even if he/she contributed only one PK parameter value to the statistical assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol / Liter
Arm/Group | 100 mg [14C]-Radiolabeled BI 1358894 (Part 1)
Number analyzed (Participants) | 8
nanomol / Liter
  BI 1358894 | 657 (43.2)
  [14C] BI 1358894-EQ | 2070 (28.4)

4. Secondary Outcome: Part 2: Area Under the Concentration-time Curve of Non-radiolabeled BI 1358894 in Plasma Over the Time Interval From 0 to 24 (AUC0-24)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 24 hours(AUC0-24) was determined for non-radiolabeled BI 1358894.
Time Frame: At 2 hours (h) before first drug administration and at 30 minutes (min), 1h, 2h, 4h, 5h, 6h, 7h, 8h, 10h, 12h, 14h and 24h after first drug administration.
Population: Pharmacokinetic set (PKS) Part 2: This subject set included all subjects in the TS who provided at least one primary or secondary PK parameter that was not excluded according to the description above. Thus, a subject was included in the PKS, even if he/she contributed only one PK parameter value to the statistical assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanomol / Liter
Groups:
- 100 mg BI 1358894 (Part 2): Multiple doses (MD) of 2 non-radiolabelled film-coated tablets of 50 milligram (mg) BI 1358894 were administered orally once daily (QD) from Day 1 to Day 21 with 240 milliliter (mL) of water .
Arm/Group | 100 mg BI 1358894 (Part 2)
Number analyzed (Participants) | 7
Hours*nanomol / Liter | 5200 (20.1)

5. Secondary Outcome: Part 2: Maximum Measured Concentration of Non-radiolabeled BI 1358894 in Plasma (Cmax)
Description: Maximum measured concentration of the analyte in plasma (Cmax) was determined for non-radiolabeled BI 1358894.
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol / Liter
Arm/Group | 100 mg BI 1358894 (Part 2)
Number analyzed (Participants) | 7
nanomol / Liter | 551 (39.1)

6. Secondary Outcome: Part 2: Area Under the Concentration-time Curve of Non-radiolabeled BI 1358894 in Plasma at Steady State Over a Uniform Dosing Interval τ (AUCτ,ss)
Description: Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) was determined for non-radiolabeled BI 1358894. Tau = 24 hours.
Time Frame: At 480h, 480.5h, 481h, 482h, 484h, 485h, 486h, 487h,488h, 490h, 492h, 494h and 504h after first drug administration.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours * nanomol / Liter
Arm/Group | 100 mg BI 1358894 (Part 2)
Number analyzed (Participants) | 7
Hours * nanomol / Liter | 14400 (11.1)

7. Secondary Outcome: Part 2: Maximum Measured Concentration of Non-radiolabeled BI 1358894 in Plasma at Steady State Over a Uniform Dosing Interval τ (Cmax,ss)
Description: Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmax,ss) was determined for non-radiolabeled BI 1358894. Tau = 24 hours.
Time Frame: At 480h, 480.5h, 481h, 482h, 484h, 485h, 486h, 487h,488h, 490h, 492h, 494h and 504h after first drug administration.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol / Liter
Arm/Group | 100 mg BI 1358894 (Part 2)
Number analyzed (Participants) | 7
nanomol / Liter | 1030 (16.5)

ADVERSE EVENTS:
Time Frame: For all AEs, including all-cause mortality: From first drug administration until end of trial, up to 50 days for part 1 and up to 62 days for part 2.
Description: Treated Set (TS): This subject set included all subjects who entered the study who were documented to have received at least one dose of study drug.
Arm/Group | 100 mg [14C]-Radiolabeled BI 1358894 (Part 1) | 100 mg BI 1358894 (Part 2)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 5/8 | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg [14C]-Radiolabeled BI 1358894 (Part 1) (N=8) | 100 mg BI 1358894 (Part 2) (N=7)
Catheter site irritation (General disorders) | 0 | 3
Vessel puncture site haematoma (General disorders) | 0 | 2
Catheter site haematoma (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Medical device site irritation (General disorders) | 0 | 1
Catheter site erythema (General disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Vessel puncture site pain (General disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Lip dry (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 1
Dizziness (Nervous system disorders) | 1 | 1
Head discomfort (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT04567316/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT04567316/SAP_001.pdf